CLINICAL TRIAL: NCT03076008
Title: The Impact of Tibial Tubercle-trochlear Groove Distance and Patellar Height on the Outcome of Isolated Medial Patellofemoral Ligament Reconstruction
Acronym: TT-TG Outcome
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: International Society of Arthroscopy, Knee Surgery and Orthopaedic Sports Medicine (Unknown); Ohio State University (Other); OrthoSport Victoria (Unknown)
Responsible Party: Sponsor
Other Study IDs: ORSU-2019-27540
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Patellar Dislocation
MeSH Terms: conditions — Patellar Dislocation | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MPFL Reconstruction: Subjects undergoing MPFL Reconstruction
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No intervention

SUMMARY:
The investigators plan to perform a prospective observational cohort study of patients undergoing MPFL reconstruction for the treatment of episodic patellar instability in the absence of significant degenerative disease. The investigators will follow these study subjects for a minimum of two years to monitor their functional and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* MPFL Reconstruction

Exclusion Criteria:

* Trochleoplasty Required
* Prior ipsilateral knee surgery
* Iwano grade 2+
* CHondral injury requiring surgical treatment beyond debridement
* Major ligamentous injury to the knee

Ages: 13 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing MPFL reconstruction for patella instability
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrent Dislocation | 2 years
  Recurrent Dislocation

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Arendt, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are currently undecided